CLINICAL TRIAL: NCT04734405
Title: Phase IIb/III Parallel-arm, Random., Active-controlled, Double-blind, Double-dummy, Multicenter, Non-inferiority Study in Patients With RVVC to Compare Efficacy, Safety and Tolerability of Topically Administered ProF-001 to Oral Fluconazole
Brief Title: A Phase IIb/III Study of Prof-001 for the Treatment of Patients With Recurrent Vulvovaginal Candidiasis (RVVC)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ProFem GmbH (Industry)
Collaborators: Montavit Ges.m.b.H. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ProF-001 IIb-III
Record Dates: First submitted 2020-11-30; First posted 2021-02-02 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Vulvovaginal Candidiasis
Keywords: Recurrent VVC; RVVC; Vulvovaginal candidiasis; ProF-001; Fluconazole; Vulvovaginitis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Vulvovaginitis | interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: Parallel-arm, Randomized, Active-controlled, Double-blind, Double-dummy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProF-001 Group (Experimental): ProF-001 Group:
  • During induction period: app. 5 g of ProF-001 for 6 days (twice daily app. 2.5 g vulvar/ intravaginal application of cream), followed by 4 days of app. 2.5 g of ProF-001 at bedtime and 1 placebo capsule on days 1, 4, and 7 and
  • During maintenance period: 2 doses of app. 2.5 g of ProF-001 per week for 22 weeks (total of 44 single doses) and 1 placebo capsule per week for 24 weeks
  Interventions: Drug: Prof-001; Drug: Placebo capsule
- Fluconazole Group (Active Comparator): Fluconazole Group:
  * During induction period:
    1 Fluconazole 150 mg capsule on days 1, 4, and 7 and a daily dose of app. 5 g of placebo cream for 6 days (twice daily 2.5 g vulvar/ intravaginal application of cream), followed by 4 days of 2.5 g of placebo cream at bedtime and
  * During maintenance period:
    1. capsule of fluconazole 150 mg per week for 24 weeks and two doses of 2.5 g of placebo cream per week for 22 weeks (total of 44 single doses)
  Interventions: Drug: Fluconazole 150 mg; Drug: Placebo cream

INTERVENTIONS:
Drug: Prof-001 — Prof-001 cream
  Arms: ProF-001 Group
Drug: Fluconazole 150 mg — Fluconazole capsule
  Arms: Fluconazole Group
Drug: Placebo cream — ointment base to mimic Prof-001
  Arms: Fluconazole Group
Drug: Placebo capsule — encapsulated lactose powder to mimic 150 mg fluconazole capsule
  Arms: ProF-001 Group

SUMMARY:
This is a prospective, randomized, multi-center, active-controlled, double-blind, double-dummy, multicenter, non-inferiority study comparing the clinical efficacy, safety and tolerability of ProF-001 to fluconazole.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 1:1 ratio to receive either ProF-001 or fluconazole for the treatment of RVVC.

Patients diagnosed with RVVC will be randomized to either ProF-001 or fluconazole treatment. Treatment schedule will start with an induction period of 10 (+4) days followed by a six months maintenance period and a subsequent 6 months follow-up (observation) period after end of active treatment.

Any episode of VVC grade > = 3 and positive vaginal smear (native or KOH) with budding yeasts, pseudohyphae or hyphae from test of cure (TOC) visit onwards will be considered as relapse of VVC.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years
* Patients suffering from an acute episode in RVVC, characterized by:
* Positive vaginal smear (native or KOH) for budding yeasts and/or (pseudo-) hyphae, normal or intermediate flora
* Two or more of the following signs and symptoms of VVC that are characterized as moderate or severe: itching, burning, irritation, edema, redness, or excoriation/fissure (Table 2).
* At least 3 previous episodes of VVC during the last 12 months (i.e. at least 4 episodes including the current episode)
* Readiness for sexual abstinence from start of treatment until test of cure (TOC) - visit
* Ability to understand trial instructions and rating scales as well as ability to comply with treatment
* Written informed consent

Exclusion Criteria:

* Known hypersensitivity to clotrimazole, diclofenac, fluconazole or any other ingredient of the investigational medicinal product
* Pregnancy or breast feeding at time of screening (for all females of childbearing potential, negative pregnancy test at screening and monthly during active treatment period will be performed). Females in childbearing potential must use adequate contraception during the active treatment period (sexual abstinence is an accepted method of birth control)
* Menstrual bleeding (spotting is not an exclusion criterion) during the first three days of treatment during the induction period
* Acute cystitis diagnosed by anamnesis and urinary dip stick (positive for leukocytes and nitrites) during screening examination
* Patients with other infectious causes of vulvovaginitis assessed during gynecological examination at screening (e.g., bacterial vaginosis, Trichomonas vaginalis, Herpes simplex)
* Patients with other clinical gynecological abnormalities, such as infections of the upper urogenital tract (pelvic inflammatory disease, adnexitis) or known high-grade cervical dysplasia at screening
* Subjects with another vaginal or vulvar condition that would confound the interpretation of clinical response (e.g. lichen sclerosus, neuropathic pain, herpes zoster)
* Treatment with antimycotics (systemic or vaginal) within the prior 3 days of randomization or during study period other than IMP (investigational medicinal product)
* Chronic (daily) use of non-steroidal anti-inflammatory medication during induction and maintenance period (>4 weeks)
* Vaginal or oral antibiotic treatment during induction period
* Vaginal use of corticosteroids, chronic systemic (oral, rectal or intravenous) use of corticosteroids during treatment and follow-up period (≥ 5 mg oral prednisolone/d or equivalent dose > 4 weeks). Topical dermal (except vulvar), intranasal or inhalative corticosteroids for allergy, asthma or chronic obstructive pulmonary disease allowed.
* Vaginal use of antihistaminic drugs during induction period
* Patients receiving anti-estrogen treatment for breast cancer, patients receiving immunosuppressive drugs
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption."
* Active malignancy (except non-melanoma skin cancer, or carcinoma in situ of cervix) or current treatment with anticancer therapy (chemotherapy, immunotherapy, radiotherapy, hormone therapy for cancer treatment, targeted therapy or gene therapy)
* Known major uncontrolled medical disorder(s) that renders the subject unsuitable for participation in the study, including but not limited to: comorbid condition with an estimated life expectancy of ≤ 12 months, known acquired immune deficiency syndrome, patients with chronic kidney disease on dialysis, patients with severe pulmonary (requiring home oxygen, uncontrolled COPD (chronic obstructive pulmonary disease) Gold III/ IV) or cardiovascular conditions (heart failure NYHA IV)
* Participation in another interventional clinical trial within the last 30 days
* Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse) or relationship to the sponsor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with at least one episode of clinical relapse of VVC during the 12 months study period. | after 12 months
  Registration of the number of patients with a clinical relapse within 12 months after randomization, clinical relapse of VVC is defined as severity score of VVC grade ≥ 3 with positive vaginal smear (native or KOH) with budding yeast or hyphae)

SECONDARY OUTCOMES:
Proportion of patients with clinical cure (absence of signs and symptoms of VVC) at 6, 8, 10 and 12 months after randomization | 6, 8, 10, 12 months
  Registration of the number of clinically cured patients throughout the study period by determination of severity score values.
Percentage of patients with clinical cure (defined as absence of signs and symptoms of VVC) at the test of cure visit, day 10 (+ 4 days) | after 2 weeks
  Registration of patients with a severity score value of 0 after therapy of the acute phase at TOC visit
Patient reported outcome of time to termination of clinical symptoms using the 11-point numeric rating scale (NRS) for burning, itching, soreness/irritation | within 2 weeks after randomization
  Registration of duration of the acute episode by decrease of NRS values in a self-assessment tool, reported in a paper diary or an electronic patient reported outcome (ePRO) system
Symptom relief reported by patients within the first 6 to 12 hours and following day after first application. Symptom relief as improvement of ≥ 2 points of symptoms compared to pre-treatment in the NRS. | 48 hours
  Registration of rapid pain release by a patient reported outcome tool by measuring the decrease of NRS values for burning, itching, soreness/irritation

OTHER OUTCOMES:
Improvement of patient reported health related quality of life score at the end of the observation period using the EQ-5D questionnaire | 0, 6 and12 months
  Registration of changes of health related quality of life (HRQoL)- score values at 0, 6 and 12 months
Sexual function related to pain and improvement thereof (see Annex I) | 0, 6 and12 months
  Evaluation of sexual function by changes of score values in a questionnaire regarding sexual function after 0, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kiss, Prof., Principal Investigator — Universitätsklinik für Frauenheilkunde
Locations (29):
- Austria (7):
  - Ordination Dr. Nehoda, Innsbruck, Tyrol
  - Ordination Dr. Peter Brock, Innsbruck, Tyrol
  - Universitätsklinik für Gynäkologie und Geburthilfe, Uni-Klinik IBK, Innsbruck, Tyrol
  - Ordination Dr. Mayr, Kufstein, Tyrol
  - Ordination Dr. Fischer, Bregenz, Vorarlberg
  - Universitätsklinik für Frauenheilkunde, AKH, Vienna
  - Ambulatorium für Pilzinfektionen und andere infektiöse venero-dermatologische Erkrankungen, Vienna
- Poland (13):
  - Provita Sp. z o.o. Fabryczna 13 D, Katowice
  - CMR, Katowice
  - Centrum Zdrowia Kobiety Komed,, Kielce
  - Komed, Kielce
  - PZS Oleśnica, Oleśnica
  - Fem-Med, Poznan
  - Gaja Poradnie Lekarskie, Poznan
  - Bonus 2001 Sp. z o.o. Sp. K., Skórzewo
  - Gabinety Lekarskie SIGNUM, Skórzewo
  - DC-MED., Dworcowa 5, Swidnica
  - Astimed Sp. z o.o.,, Warsaw
  - Centrum medyczne Lux MED, Warsaw
  - Centrum Medyczne LUX MED Swidnicka 40, Wroclaw
- Slovakia (9):
  - BESME s.r.o, Bánovce nad Bebravou
  - MILLY s.r.o., Bratislava
  - Gynedur s.r.o., Dubnica nad Váhom
  - MCM GYNPED s.r.o., Dubnica nad Váhom
  - Gyncentrum Nitra s.r.o., Nitra
  - GYNAMA s.r.o., Nové Mesto nad Váhom
  - BrenCare s.r.o, Poprad
  - GYNECARE s.r.o., Púchov
  - Gyneka s.r.o., Privatna gynekologicko porodnicka ambulancia, Trenčín

IPD SHARING:
Plan to Share IPD: No